CLINICAL TRIAL: NCT06612892
Title: Immersive Versus Passive Virtual Reality on Upper Limb Pain and Range of Motion in Pediatric Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haytham Mostafa, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Haitham-005156
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Virtual Reality; Immersive Virtual Reality; Pediatric Burn; Passive Virtual Reality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality (Experimental): consisted of 30 patients and received procedure as immersive virtual reality program selected to enhance patient to use his upper limbs in order to interact with the show or game selected
  Interventions: Device: Virtual reality games in immersive VR modality; Other: traditional physiotherapy
- Passive virtual reality (Active Comparator): consisted of 3o patients and received procedure as passive virtual reality program as the patient just wear the headset with a view or show meant only to distract pain while following therapist commands to do active or active assisted upper limbs ROM ex.
  Interventions: Device: Virtual reality show in passive VR modality:; Other: traditional physiotherapy

INTERVENTIONS:
Device: Virtual reality games in immersive VR modality — virtual reality involved three characters: a muscular boxer, a superhero, and a rock climber, with patients performing tasks in standing or sitting. Each experience takes 6 minutes, with 5-minute intervals between. Experimenters will instruct users on hand controls and virtual body observation.
  Arms: Immersive virtual reality
Device: Virtual reality show in passive VR modality: — In this modality the patient was asked to have a comfortable seat wearing the head set without holding the controllers , the therapist will play a relaxing show as a nature view or colorful scene as a sort of relaxation and mind distraction for around 20 minutes while asking the patient to perform upper limb muscle ROM exercise in active or active assisted form.
  Arms: Passive virtual reality
Other: traditional physiotherapy — Includes stretching exercise for upper limb muscles affected by burn, scar tissue release , and splinting technique.

SUMMARY:
The purpose of the present study was to declare the difference between using immersive virtual reality vs passive virtual reality on pain management and improvement of ROM post physiotherapy exercise and mobilization sessions in pediatric burn patients.

DETAILED DESCRIPTION:
Burn injuries are devastating and cause long-term damage to health. Thermal injuries, caused by hot liquids, solids, or fire, account for the majority of these injuries. Around 11 million burn cases occur annually worldwide. Rehabilitation aims to improve joint range od motion and control pain. Nonpharmocologic strategies like hypnosis and VR systems have shown promise in pain control. Multidisciplinary interventions from psychologists, physiotherapists, and pain management specialists can contribute to patient recovery. VR offers a holistic care device for pediatric burn patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty patients have 2nd degree thermal burn injury, from both genders their ages will be ranged from 7 - 17 years old.
2. They will be diagnosed by their physicians with 2nd degree thermal burn injury affecting upper limbs and referred for physical therapy management .
3. TBSA calculated up to 9 for one upper limb.
4. The patients will be in the acute stage post burn injury; the duration of burn will be 3 weeks post injury.
5. Medically and psychologically stable patients

Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

1. Cardiac diseases.
2. Hand Burn
3. Exposed tendons.
4. Patients who suffer from skin diseases, diabetes, varicose veins, and peripheral vascular diseases.
5. Patients with life threatening disorders as renal failure, myocardial infarction or other similar diseases.
6. Patients with facial burn.
7. Patients will have an inability to tolerate visual stimulation (e.g., susceptibility to migraines aggravated by light) or inability to tolerate the head mounted display (e.g., sensitivity to touch around the face and head).
8. Patients with visual or auditory disorders.
9. Patients with unstable fractures.
10. Central Nervous System (CNS) problems.
11. Patients with medical red flags as severe psychiatric disorder or cognitive deficits .
12. Medically unstable and uncooperative patients.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
assessing the pain intensity using Colored Analog Scale (CAS) | at baseline and after 6 weeks
  The Colored Analog Scale (CAS) is a thermometer-like tool that gradually darkens red as you progress, allowing children to indicate their pain levels with markers on the scale's back.
assessing the range of motion using digital goniometer | at baseline and after 6 weeks
  The physical therapist will have to measure ROM before and after the intervention to monitor the improvement ,as the study focus on upper limb range of motion , following joints movement will be measured : shoulder flexion and abduction , elbow flexion and extension , wrist flexion and extension , forearm supination and pronation)

CONTACTS AND LOCATIONS:
Locations (1):
- Haytham Mostafa Youssef, Cairo, Egypt